CLINICAL TRIAL: NCT06618144
Title: Conversational AI to Improve PeRiconception Care Access
Brief Title: Conversational Artificial Intelligence (AI) to Improve PeRiconception Care Access
Acronym: CIRCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Memora Health Inc (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OBGYN-PEACE-QI-1
Record Dates: First submitted 2024-08-21; First posted 2024-10-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Early Pregnancy Loss; Early Pregnancy
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIRCA Texting (Experimental): Participants will be invited to text with a secure, closed artificial intelligence system with clinician oversight to triage patients along predetermined algorithms related to early pregnancy care.
  Interventions: Other: Texting platform

INTERVENTIONS:
Other: Texting platform — Participants will be invited to text with a secure, closed artificial intelligence system with clinician oversight to triage patients along predetermined algorithms related to early pregnancy care.

SUMMARY:
The goal of this project, Conversational Artificial Intelligence (AI) to Improve PeRiconception Care Access (CIRCA), is to engage patients in care early in pregnancy (before prenatal care starts) and safely triage concerns to PEACE to reduce unnecessary emergency department visits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Seeking to establish care at the Hospital of the University of Pennsylvania OR seeking care in the Emergency Department or Perinatal Evaluation Center.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-09-21 (Actual); Study Completion 2025-09-21 (Actual)

PRIMARY OUTCOMES:
Time to initiating care (days) | Up to 3 months
  Time from first contact to initiating pregnancy related care

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No